CLINICAL TRIAL: NCT07004946
Title: Diagnostic Value of Confocal Laser Endomicroscopy (CelTouch) for Peripheral Lung Lesions
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, Professor, Guangzhou Medical University
Other Study IDs: CelTouch clinical trial
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Pulmonary Lesion
Keywords: peripheral pulmonary lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Confocal laser endomicroscopy group: Utilize confocal laser endomicroscopy for the examination of peripheral lung lesions in patients.

SUMMARY:
This study uses CelTouch to explore patients with lung lesions scheduled for lung biopsy. By comparing with preclinical CLE images and pathological images, CLE diagnostic criteria for benign and malignant lung lesions under the microscope will be established; the performance of CLE in diagnosing peripheral lung lesions will be validated through multicenter clinical research; and a CLE atlas for peripheral lung lesions will be constructed to establish a visual classification diagnostic system for peripheral lung lesions.

(1) Comparative Study of In Vivo CLE Images and Pathological Images in the Diagnosis of Peripheral Lung Lesions

1. Collect CLE images and histopathological sections of clearly diagnosed peripheral lung lesions.
2. A diagnostic team composed of 1 bronchoscopy expert, 1 pathology expert, and 2 CLE experts will correlate in vivo and ex vivo CLE images of lung lesions with corresponding pathological images, analyze CLE image characteristics of benign and malignant lung lesions, and establish CLE diagnostic criteria for benign and malignant lung lesions.

(2) Validation Study of the Diagnostic Performance of Confocal Laser Endomicroscopy in Peripheral Lung Lesions

1. Multicenter screening of corresponding subjects according to inclusion and exclusion criteria, collection of corresponding videos and images during surgery, and recording of observed characteristic images based on pre-established diagnostic characteristics and criteria.
2. The diagnostic team and sub-center representatives (5 in total) will perform offline interpretation of the collected images and videos, and evaluate the diagnostic performance of CLE in peripheral lung lesions using the accurate diagnostic results obtained from postoperative histopathology or 6-month clinical follow-up as the standard.
3. Establishment of a CLE Atlas and Classification System for Lung Lesions

(1) Collect large-scale in vivo and ex vivo CLE images and pathological images of clearly diagnosed lung lesions from multiple centers.

(2) Select typical in vivo and ex vivo CLE images of lung lesions with the same pathological type and corresponding pathological images, and jointly describe the CLE image diagnostic characteristics by pathology experts and CLE experts to establish a CLE atlas for peripheral lung lesions.

(3) Establish a visual classification system for the internal structure of peripheral lung lesions based on the special signs in CLE images of lung lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years, with lung lesions detected by chest CT and scheduled for lung biopsy;
2. Preoperative CT indicates the presence of a bronchus leading to the lesion to be biopsied;
3. Able to understand and willing to sign a written informed consent form. -

Exclusion Criteria:

1. Those with contraindications to general anesthesia or bronchoscopy;
2. Patients with uncorrectable coagulation disorders;
3. Unable to discontinue therapeutic anticoagulants within an appropriate time interval before surgery;
4. Patients with severe liver or kidney dysfunction, cardiovascular and cerebrovascular diseases, mental illnesses, etc.;
5. Pregnant or lactating patients;
6. Those without a clear histological or clinical diagnosis;
7. Subjects deemed unsuitable by the investigator. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. All subjects have completed CelTouch examination
  2. Each subject has obtained a clear histological diagnosis or clinical follow-up diagnosis for 6 months
Sampling Method: Non-Probability Sample
Enrollment: 286 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 6 months after procedure
  diagnostic yield=(The number of cases with a definitive diagnosis / The total number of cases enrolled in the trial) × 100%

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong 510163, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wijmans L, Yared J, de Bruin DM, Meijer SL, Baas P, Bonta PI, Annema JT. Needle-based confocal laser endomicroscopy for real-time diagnosing and staging of lung cancer. Eur Respir J. 2019 Jun 20;53(6):1801520. doi: 10.1183/13993003.01520-2018. Print 2019 Jun. PMID 31023849